CLINICAL TRIAL: NCT03128879
Title: A Phase II Study of Venetoclax (ABT-199) Consolidation for Patients Currently Receiving Ibrutinib or Acalabrutinib for High-risk CLL
Brief Title: Venetoclax With Ibrutinib or Acalabrutinib in Pts. With High-risk CLL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0785; NCI-2018-01182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0785 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ibrutinib, acalabarutinib) (Experimental): Patients receive venetoclax PO QD and ibrutinib PO QD and acalabrutinib PO BID. Treatment repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Acalabrutinib — Given BID

SUMMARY:
This is a single center, open-label, phase II study of venetoclax (ABT-199) added to ibrutinib or acalabrutinib in patients with high-risk CLL who have received at least 12 months of ibrutinib or acalabrutinib monotherapy.

The study will estimate the therapeutic efficacy of venetoclax consolidation in patients who have detectable CLL after receiving ibrutinib or acalabrutinib for at least 12 months and who have high risk CLL.

DETAILED DESCRIPTION:
Primary Objective:

1. To estimate the therapeutic efficacy of venetoclax consolidation in patients who have detectable CLL after receiving ibrutinib or acalabrutinib for at least 12 months and who have high risk CLL. High risk is defined as the presence of at least one of: del(17p); TP53 mutation; complex metaphase karyotype; patients who have developed mutations in BTK and/or PLCG2, will be eligible if they have no clinical or laboratory evidence of progressive disease. The primary endpoint will be the rate of MRD-negativity in the bone marrow, using an assay method with at least 0.01% sensitivity after 12 cycles of combination therapy. One cycle is 4 weeks of treatment.

Secondary Objectives:

1. Determine CR/CRi rate after 6, 12 18 and 24 cycles of combination therapy, in patients who were not in CR/Cri at study initiation and estimate the time to best response with this combination.
2. Determine the cumulative rate of bone marrow minimal residual disease (MRD)-free complete responders by an assay method with at least 0.01% sensitivity and median time to MRD-negativity.
3. Determine the safety of combined ibrutinib and venetoclax.
4. Determine the progression-free and overall survival.

OUTLINE: This is a dose-escalation study of venetoclax.

Patients receive venetoclax orally (PO) once daily (QD) and ibrutinib PO QD and acalabrutinib PO BID. Treatment repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of CLL/CLL and have high-risk cytogenetic features or molecular features, defined as: del(17p), mutated TP53, complex metaphase karyotype (defined as 3 unrelated chromosomal abnormalities, present in at least 2 metaphases on conventional, stimulated cytogenetic analysis)

   *** Note: some patients treated with ibrutinib or acalabrutinib may no longer have detectable FISH, karyotypic or molecular abnormalities after 12 months of therapy. These patients will be eligible if they fulfill the above criteria on a bone marrow biopsy or peripheral blood specimen taken either prior to starting ibrutinib or acalabrutinib, provided they did not receive treatment for their CLL between the date of the lab test and starting ibrutinib or acalabrutinib or at some time during their ibrutinib therapy and analyzed at a CLIA-accredited laboratory.
2. Patients must have received at least 12 months of ibrutinib or acalabrutinib therapy and have measurable CLL by at least one of the following:

   * Absolute monoclonal lymphocyte count > 4000/L; OR
   * Measurable lymph nodes with at least one node >1.5 cm in diameter on CT; OR
   * Bone marrow with >/= 30% lymphocytes on aspirate differential OR
   * Detectable CLL cells using a standardized flow cytometry assay for minimal residual disease
3. Age 18 years or older.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
5. Patients must have adequate renal and hepatic function:

   * Serum bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for patients with Gilbert's disease.
   * Serum creatinine clearance of 50ml/min (calculated or measured).
   * ALT and AST ≤3.0 x ULN, unless clearly due to disease involvement.
6. Adequate bone marrow function:

   * Platelet count of greater than 50,000/µl, with no platelet transfusion in prior 2 weeks.
   * ANC ≥1000/µl in the absence of growth factor support unless due to compromised bone marrow production from CLL, indicated by 80% CLL in marrow.
   * Hemoglobin ≥8mg/dL.
7. INR <1.5.
8. Adequate cardiac function, as assessed by:

   * Absence of uncontrolled cardiac arrhythmia.
   * Echocardiogram demonstrating LVEF ≥35%.
   * NYHA functional class ≤2.
9. Ability to provide informed consent and adhere to the required follow-up.
10. Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use use both a highly effective method of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence , or sterilized partner) and a barrier method (eg., condoms, vaginal ring, sponge, etc) during the period of therapy and for 30 days after the last dose of study drug. Women of non-childbearing potential are those who are postmenopausal (defined as absence of menses for ≥1 year) or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use effective contraception, defined above, during the study and for 30 days following the last dose of study drug.
11. Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

1. Richter transformation.
2. Active malignancy requiring systemic therapy, other than CLL, with the exception of: adequately treated in situ carcinoma of the cervix uteri; adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
3. Major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 3 weeks prior to the first dose of the study drug.
4. Grade 3 or 4 hemorrhage within the past 3 weeks.
5. Uncontrolled active infections (viral, bacterial, and fungal).
6. Females who are pregnant or lactating.
7. Known positive serology for human immunodeficiency virus (HIV).
8. Active hepatitis B infection (defined as the presence of detectable HBV DNA or HBe antigen). Patients who are HBsAg positive or HBcAb positive are eligible, provided HBV DNA is negative. These patients will have monthly monitoring of HBV DNA for the duration of the study, if clinically indicated. Please note that patients who have received IVIG may have false positive HBcAb results. In such patients, if HBV DNA and HBsAg are negative, serial HBV DNA monitoring is not necessary.
9. Active hepatitis C, defined by the detection of hepatitis C RNA in plasma by PCR.
10. Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy >20mg prednisone daily or equivalent, within 7 days of starting venetoclax.
11. Received other investigational therapeutic agent for CLL/SLL within 21 days of starting venetoclax.
12. Concurrent use of warfarin.
13. Received strong CYP3A inhibitors or strong CYP3A inducers within 7 days of starting venetoclax.
14. Consuming grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting venetoclax.
15. Prior treatment with venetoclax or other Bcl-2 inhibitor.
16. Malabsorption syndrome or other condition that precludes enteral route of administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the rate of MRD-negativity in the bone marrow, using an assay method with at least 0.01% sensitivity after 12 cycles of combination therapy. One cycle is 4 weeks of treatment. | through study completion, an average of 1 year
  One cycle is 4 weeks of treatment. (each cycle 28 days)

SECONDARY OUTCOMES:
Determine complete remission CR/complete remission with incomplete hematologic recovery CRi rate of combination therapy in patients who were not in CR/Cri at study initiation and estimate the time to best response with this combination. | through study completion, an average of 1 year
  after 6, 12, 18 and 24 cycles (each cycle 28 days)
Determine the cumulative rate of bone marrow minimal residual disease (MRD)-free complete responders by an assay method with at least 0.01% sensitivity and median time to MRD-negativity. | through study completion, an average of 1 year
Determine the safety of combined ibrutinib and venetoclax. | through study completion, an average of 1 year
  Safety data will be summarized by category, severity and frequency. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval. The severity of the toxicities will be graded according to the NCI CTCAE v4.0 whenever possible.
Determine the progression-free survival | through study completion, an average of 1 year
Determine the overall survival. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org